CLINICAL TRIAL: NCT06078527
Title: Assessment of Laryngopharyngeal Sensation in Patients With Laryngopharyngeal Disorders
Brief Title: Assessment of Laryngopharyngeal Sensation: Cancer Survivor Cohort
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Spasmodic Dysphonia Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 232011; NCI-2023-10667 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2023-10-05; First posted 2023-10-12 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Presbylarynx; Aspiration; Spasmodic Dysphonia; Globus Pharyngeus; Larynx Paralysis; Laryngeal Disease; Vocal Cord Paralysis; Iatrogenic Injury; Sensory Neuropathy
Keywords: Cancer survivors; Previous cancer treatment; Laryngopharyngeal disorders
MeSH Terms: conditions — Dysphonia; Globus Sensation; Vocal Cord Paralysis; Laryngeal Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Cancer Survivors (Experimental): Participants will attend a single 15-30 minute study session during which they will answer questionnaires (5-10 minutes) and undergo laryngopharyngeal sensory testing (10-20 minutes). There will be up to 2 years of medical record follow up after completing the main study.
  Interventions: Device: Cheung-Bearelly Aesthesiometer; Procedure: Transnasal Laryngoscopy; Other: Questionnaires

INTERVENTIONS:
Device: Cheung-Bearelly Aesthesiometer — The Cheung-Bearelly Aesthesiometer will be used to deliver a range of calibrated stimuli through the channeled flexible laryngoscope to assess sensation of the laryngopharynx.
  Other Names: Aesthesiometer
Procedure: Transnasal Laryngoscopy — A procedure to examine your larynx (voice box)
  Other Names: Transnasal Flexible Laryngoscopy
Other: Questionnaires — Patient-reported health and behavioral outcomes measures will be administered

SUMMARY:
A previous study completed in 2022 (NCT05158179) was conducted using cohorts of healthy controls, and adults with general laryngopharyngeal disorders. This study will expand on the previous research to include a separate cohort of adults being seen in clinic for an existing laryngopharyngeal disorder resulting from previous radiation or other cancer treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Laryngeal sensation as measured by elicitation of laryngeal adductor reflex (LAR).

II. To compare the elicitation of laryngeal adductor reflex (LAR) threshold/probability to the Penetration-Aspiration Scale (PAS).

SECONDARY OBJECTIVES:

I. To assess patient-reported laryngeal sensation (PRLS) following stimulus and perceptual strength.

II. To assess laryngopharyngeal responses (e.g., cough, gag, swallow) following stimulus.

III. To assess patient reported outcomes (PROs).

EXPLORATORY OBJECTIVES:

I. To compare the elicitation of laryngeal adductor reflex (LAR) threshold/probability to:

* modified barium swallow (MBS) study kinematics;
* MBS Dynamic Imaging Grade of Swallowing Toxicity (MBS DIGEST);
* MD Anderson Dysphagia Inventory patient reported outcomes measure (MDADI PROMs);
* Dynamic Imaging Grade of Swallowing Toxicity for Flexible Endoscopic Evaluation of Swallowing (DIGEST-FEES)
* Flexible Endoscopic Evaluation of Swallowing Visual Analysis of Swallowing Efficiency and Safety (FEES VASES).

OUTLINE:

Participants receiving care at University of California, San Francisco (UCSF) for an existing laryngopharyngeal disorder resulting from previous radiation or other cancer treatments will undergo laryngopharyngeal sensory testing at a single visit. There will be up to 2 years of medical record follow up after completing the main study. Data collected from this separate cohort may be compared with historical data collected in a previous study (NCT05158179).

ELIGIBILITY:
Inclusion Criteria:

1. Age <=18 years.
2. Individuals without a laryngopharyngeal disorder (health controls) or with a laryngopharyngeal disorder. Laryngopharyngeal disorder includes but is not limited to: presbylarynx, aspiration; spasmodic dysphonia; globus pharynges; vocal fold paralysis; iatrogenic injury to the larynx; muscle tension dysphonia; neurogenic dysphagia; laryngeal sensory neuropathy; and laryngopharyngeal disorders resulting from prior radiation therapy in individuals with a history of head and neck cancer who have completed radiation therapy as primary or adjuvant cancer treatment
3. Ability and willingness to comply with study procedures.
4. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Non-English speaking.
2. Laryngopharyngeal structures are not accessible on exam.
3. Known contraindication to any study-related procedure, or history of being unable to tolerate laryngoscopy.
4. Vocal fold immobility or severe hypomobility on adduction.
5. For head and neck cancer survivors only: Currently undergoing radiation therapy for head and neck cancer (i.e., primary/adjuvant radiation therapy treatment plan is not yet completed).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with triggered/positive laryngeal adduction response (LAR) | 1 day
  Elicitation of LAR is defined as a unilateral or bilateral laryngeal adduction immediately following laryngeal stimulus through frame-by-frame analysis of video recordings (visualized on laryngoscopy). An acceptable tactile stimulus is near orthogonal (less than 30 degrees deviation) to the mucosal surface and unobstructed by salivary forces. The percentage of participants with LAR will be reported
Median scores on the Penetration-Aspiration Scale (PAS) | 1 day
  The PAS is a widely-used ordinal scale metric used to describe severity of aspiration. The PAS score is multidimensional, i.e., include several observations within each score: (1) depth of airway invasion (material above, contacting, or below the level of vocal folds; (2) whether or not there is material remaining after the swallow (ejected, not ejected); and (3) the patient's response to material present in the airway (effort to clear the material). The PAS is an 8-point ordinal scale, with a total score ranging from 1 representing the least and 8 representing the highest or most severe score.

SECONDARY OUTCOMES:
Median scores on the participant-reported laryngeal sensation (PRLS) | 1 day
  The PRLS is defined as a binary response to participants' self-reported detection of laryngeal stimulation. Once the participant indicates they perceived the stimulus, the research team will ask the participant to provide a perceptual strength rating on a 1-10 scale, with higher scores indicated a greater strength of stimulus.
Percentage of participants with visualized laryngopharyngeal responses | 1 day
  Percentage of participants with visualized laryngopharyngeal responses (e.g., cough, gag, swallow) following stimulus will be recorded by the clinician and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Yue Ma, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No